CLINICAL TRIAL: NCT03456362
Title: Promoting Motor Recovery in Patients With Stroke by Enhancing Cerebellar-cortical Plasticity: a Randomized Double Blinded Controlled Repetitive TMS Trial
Brief Title: Cerebellar rTMS to Improve Gait Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Giacomo Koch, Head of Laboratory, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2011-02349953
Record Dates: First submitted 2018-02-19; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Gait, Hemiplegic
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebellar iTBS (Active Comparator): Intermittent theta burst stimulation applied immediately before the daily physical therapy session for a period of three weeks.
  Interventions: Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION
- Sham iTBS (Sham Comparator): Sham intermittent theta burst stimulation applied immediately before the daily physical therapy session for a period of three weeks.
  Interventions: Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION

INTERVENTIONS:
Device: REPETITIVE TRANSCRANIAL MAGNETIC STIMULATION — theta burst stimulation (TBS) is a novel form of repetitive transcranial magnetic stimulation that mimics protocols inducing long-term potentiation (LTP) or long-term depression (LTD) in animal models. Whereas continuous TBS (cTBS) induces long-lasting inhibition of cortical areas, iTBS exerts the opposite effect, increasing cerebellar excitability

SUMMARY:
The cerebellum is known to be strongly implicated in the functional reorganization of motor networks in stroke patients, especially for gait an balance functions. Repetitive transcranial magnetic stimulation of the cerebellum can be used to enhance these adaptive processes in stroke recovery. In this randomized, double blind, sham-controlled trial we aim to investigate the efficacy and safety of cerebellar intermittent theta burst stimulation coupled with intensive physical therapy in promoting gait recovery in hemiparetic patients due to recent stroke in the territory of the contralateral middle cerebral artery

ELIGIBILITY:
Inclusion Criteria:

* First ever-chronic ischemic stroke, i.e. at least 6 months after the stroke event,
* Left or right subcortical or cortical lesion of the middle cerebral artery with medium-severity stroke NHISS <15 (All lesions must be documented by magnetic resonance imaging (T1- and T2-weighted images; 1.5T, GE scanners)
* No contraindication to brain MRI
* MEP recordable in order to evaluate the resting motor threshold (RMT)

Exclusion Criteria:

* Epilepsy
* Severe general impairment or concomitant diseases (tumors, etc.)
* Age> 80 years
* Infections in progress
* Patients with neurological diseases beyond stroke or with neuropsychiatric disorders or with neuropsychological disorders that could potentially compromise informed consent or compliance during the study.
* Treatment with benzodiazepines, baclofen, antidepressants, clonidine, beta blockers and other potentially interfering drug treatments on plasticity phenomena.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) for gait and balance | Change from baseline at the end of three weeks treatment
  Assessment of gait and balance functions

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA) scale | Change from baseline at the end of three weeks treatment
  Assessment of motor functions
Barthel Index (BI) | Change from baseline at the end of three weeks treatment
  Assessment of functional abilities
Neurophysiological assessment of cortical activity | Change from baseline at the end of three weeks treatment
  evaluation of cortical activity by means of TMS in combination with EEG
Gait analysis | Change from baseline at the end of three weeks treatment
  evaluation of locomotion

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Lucia Foundation, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koch G, Bonni S, Casula EP, Iosa M, Paolucci S, Pellicciari MC, Cinnera AM, Ponzo V, Maiella M, Picazio S, Sallustio F, Caltagirone C. Effect of Cerebellar Stimulation on Gait and Balance Recovery in Patients With Hemiparetic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Feb 1;76(2):170-178. doi: 10.1001/jamaneurol.2018.3639. PMID 30476999